CLINICAL TRIAL: NCT07174453
Title: A Late Phase Randomized Open-Label Multi Cohort Trial to Evaluate irAEs With Different Standard of Care Dosing Strategies of Standard of Care Immunotherapies
Brief Title: Trial to Evaluate irAEs With Different Standard of Care Dosing Strategies of Standard of Care Immunotherapies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Anup Kasi, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161901
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Malignancies
Keywords: Immunotherapy
MeSH Terms: interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): Pembrolizumab Cohort- Dose: 200 mg Route: IV Schedule: Once every 3 weeks Overall Treatment Duration per Participation: Average of 12 months Cycle Length: Per SOC (3 weeks)
  Nivolumab Cohort- Dose: 240 mg Route: IV Schedule: Once every 2 weeks Overall Treatment Duration per Participation: Average of 12 months Cycle Length: Per SOC (2 weeks)
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab
- Arm 2 (Experimental): Nivolumab Cohort- Dose: 480 mg Route: IV Schedule: Once every 4 weeks Overall Treatment Duration per Participant: Average of 12 months Cycle length: Per SOC (4 weeks)
  Pembrolizumab Cohort- Dose: 400 mg Route: IV Schedule: Once every 6 weeks Overall Treatment Duration per Participant: Average of 12 months Cycle length: Per SOC (6 weeks)
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nivolumab — Immunotherapy
  Other Names: Opdivo
Drug: Pembrolizumab — Immunotherapy
  Other Names: Keytruda

SUMMARY:
Phase 3/4 open label, randomized two cohort study (2 arms in each cohort).

It is hypothesized that for people with a histologically or cytologically confirmed diagnosis of malignancy, the higher dose immunotherapy (every 6 weeks Pembrolizumab 400mg dose and every 4 weeks Nivolumab 480mg dose) has more immune-related adverse events irAEs compared to lower dose (every 3 weeks Pembrolizumab 200mg dose and every 2 weeks Nivolumab 240mg dose).

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant to understand this study, and participant willingness to sign a written informed consent.
2. Males and females age ≥ 18 years
3. ECOG Performance Status (PS) 0 - 2 (Appendix A.)
4. Females of childbearing potential must have a negative urine pregnancy test 72 hours prior to initiating treatment.
5. Histologically or cytologically confirmed diagnosis of solid tumor malignancy
6. Eligible to receive pembrolizumab or nivolumab based therapy
7. Any disease setting (neoadjuvant, adjuvant, unresectable, metastatic) or any line of therapy is allowed. NOTE: Standard of care combination agents(chemotherapy, targeted therapy, biologics) are allowed because irAEs are the primary objective
8. Adequate organ function, defined as follows:

Leukocytes (White Blood Cell [WBC]) >1.0 K/UL Absolute Neutrophil Count >1.0 K/UL Platelets > 50 K/UL Hemoglobin ≥ 7 g/dL Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation Total bilirubin ≤ 1.5 x ULN Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN

Exclusion Criteria:

1. Simultaneously enrolled in any therapeutic clinical trial
2. Concurrent or planned use of other immunotherapies or radiation
3. Has not recovered from irAEs due to prior immunotherapy treatment (>=grade 2 is considered not recovered). Conditions that meet grade 2 criteria but are considered clinically stable at the discretion of the investigator will be allowed.
4. Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
5. Currently pregnant or breastfeeding
6. Has a known allergic reaction to any excipient contained in the study drug formulation
7. Active Grade 3 (per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 ) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportions of grade ≥3 immune related adverse events (irAEs) between the two arms in each cohort | 12 weeks
  Measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v 5.0

SECONDARY OUTCOMES:
All grades of immune related adverse events (irAEs) | Start of treatment to EOT. Approximate time frame 6-12 months.
  Measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Time to resolution of immune related adverse events (irAEs) | Start of treatment to end of follow up. Approximate Time Frame: 2-3 Years
  Measured by The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Time of treatment discontinuation due to immune related adverse events (irAEs) | Start of treatment to discontinuation Approximate Time Frame: 12 Months
  Duration of time from start of treatment to discontinuation, determined by medical record
Overall Response Rate (ORR) | Approximate time frame: 12 weeks
  Measured by response evaluation criteria in solid tumors (RECIST) and medical record.
Disease-Free Survival (DFS) | 6 months, 1 year, and 2 yearsApproximate time frame 3 years.
  To assess absence of disease recurrence, as determined by medical record imaging.
Progression-Free Survival (PFS) | 6 months, 1 year, and 2 yearsApproximate time frame 3 years.
  The duration of time from start of treatment until objective tumor progression or death, as determined by medical record imaging
Overall Survival (OS) | Approximate time frame: 2 years
  Duration of time from start of treatment to death, determined by medical record

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Persigehl T, Lennartz S, Schwartz LH. iRECIST: how to do it. Cancer Imaging. 2020 Jan 3;20(1):2. doi: 10.1186/s40644-019-0281-x. PMID 31900236
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER), Center for Devices and Radiological Health (CDRH), Oncology Center of Excellence (OCE). Protocol Deviations for Clinical Investigations of Drugs, Biological Products, and Devices Guidance for Industry - Draft Guidance. December 2024. Available from:https://www.fda.gov/media/184745/download . Accessed 01-21-2025
- [Background] The University of Kansas Cancer Center Clinical Trials Office Policy - Executive Resourcing Committee Submission Requirements. Version dated 08-03-2022. Cited 09-20-2024. Available from: https://kumed.sharepoint.com/sites/mykumc/cto/Documents/CTO%20Policy_ERC%20Submission.pdf#search=executive%20resource Accessed 09-20-2024
- [Background] The University of Kansas Cancer Center General Administration Guidance Document - Use of Investigator Initiated Steering Committee. Version dated 07-31-2023. Cited 09-20-2024. Available from: https://kumed.sharepoint.com/sites/mykumc/cto-training/Documents/Guidance_Use%20of%20Investigator%20Initiated%20Steering%20Committee.pdf#search=steering%20committee%20guidance%20document Accessed 09-20-2024
- [Background] European Medicines Agency. ICH Topic E 2 A Clinical Safety Data Management: Definitions and Standards for Expedited Reporting. June 1995. https://www.ema.europa.eu/en/ich-e2a-clinical-safety-data-management-definitions-standards-expedited-reporting-scientific-guideline . Cited 12-06-2024
- [Background] National Institute of Health/National Cancer Institute - Cancer Therapy Evaluation Program (CTEP). Common Terminology Criteria for Adverse Events (CTCAE). Available from: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_60 Accessed 07-05-2023.
- [Background] Bristol-Meyers Squibb Company. Nivolumab package insert revised 05-2025.
- [Background] Gritstone bio. Protocol GO-010 - A Phase 2/3, Randomized, Open-Label Study of Maintenance GRT-C901/GRT-R902, A Neoantigen Vaccine, in Combination with Immune Checkpoint Blockade for Patients with Metastatic Colorectal Cancer. Version 4.0 dated 05-31-2023.
- [Background] Ascierto PA, Del Vecchio M, Robert C, Mackiewicz A, Chiarion-Sileni V, Arance A, Lebbe C, Bastholt L, Hamid O, Rutkowski P, McNeil C, Garbe C, Loquai C, Dreno B, Thomas L, Grob JJ, Liszkay G, Nyakas M, Gutzmer R, Pikiel J, Grange F, Hoeller C, Ferraresi V, Smylie M, Schadendorf D, Mortier L, Svane IM, Hennicken D, Qureshi A, Maio M. Ipilimumab 10 mg/kg versus ipilimumab 3 mg/kg in patients with unresectable or metastatic melanoma: a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2017 May;18(5):611-622. doi: 10.1016/S1470-2045(17)30231-0. Epub 2017 Mar 27. PMID 28359784
- [Background] Puzanov I, Diab A, Abdallah K, Bingham CO 3rd, Brogdon C, Dadu R, Hamad L, Kim S, Lacouture ME, LeBoeuf NR, Lenihan D, Onofrei C, Shannon V, Sharma R, Silk AW, Skondra D, Suarez-Almazor ME, Wang Y, Wiley K, Kaufman HL, Ernstoff MS; Society for Immunotherapy of Cancer Toxicity Management Working Group. Managing toxicities associated with immune checkpoint inhibitors: consensus recommendations from the Society for Immunotherapy of Cancer (SITC) Toxicity Management Working Group. J Immunother Cancer. 2017 Nov 21;5(1):95. doi: 10.1186/s40425-017-0300-z. PMID 29162153
- [Background] Kennedy LB, Salama AKS. A review of cancer immunotherapy toxicity. CA Cancer J Clin. 2020 Mar;70(2):86-104. doi: 10.3322/caac.21596. Epub 2020 Jan 16. PMID 31944278
- [Background] ESMO. The Combination of Nivolumab and Cabozantinib Provides a New First-Line Treatment Option in Advanced Clear Cell RCC. Accessed October 22, 2021. https://www.esmo.org/oncology-news/the-combination-of-nivolumab-and-cabozantinib-provides-a-new-first-line-treatment-option-in-advanced-clear-cell-rcc
- [Background] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Background] Renner A, Burotto M, Rojas C. Immune Checkpoint Inhibitor Dosing: Can We Go Lower Without Compromising Clinical Efficacy? J Glob Oncol. 2019 Jul;5:1-5. doi: 10.1200/JGO.19.00142. PMID 31348737
- [Background] Powles T, Plimack ER, Soulieres D, Waddell T, Stus V, Gafanov R, Nosov D, Pouliot F, Melichar B, Vynnychenko I, Azevedo SJ, Borchiellini D, McDermott RS, Bedke J, Tamada S, Yin L, Chen M, Molife LR, Atkins MB, Rini BI. Pembrolizumab plus axitinib versus sunitinib monotherapy as first-line treatment of advanced renal cell carcinoma (KEYNOTE-426): extended follow-up from a randomised, open-label, phase 3 trial. Lancet Oncol. 2020 Dec;21(12):1563-1573. doi: 10.1016/S1470-2045(20)30436-8. Epub 2020 Oct 23. PMID 33284113
- [Background] Michot JM, Bigenwald C, Champiat S, Collins M, Carbonnel F, Postel-Vinay S, Berdelou A, Varga A, Bahleda R, Hollebecque A, Massard C, Fuerea A, Ribrag V, Gazzah A, Armand JP, Amellal N, Angevin E, Noel N, Boutros C, Mateus C, Robert C, Soria JC, Marabelle A, Lambotte O. Immune-related adverse events with immune checkpoint blockade: a comprehensive review. Eur J Cancer. 2016 Feb;54:139-148. doi: 10.1016/j.ejca.2015.11.016. Epub 2016 Jan 5. PMID 26765102
- [Background] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Background] Hamid O, Carvajal RD. Anti-programmed death-1 and anti-programmed death-ligand 1 antibodies in cancer therapy. Expert Opin Biol Ther. 2013 Jun;13(6):847-61. doi: 10.1517/14712598.2013.770836. Epub 2013 Feb 19. PMID 23421934
- [Background] Martins F, Sofiya L, Sykiotis GP, Lamine F, Maillard M, Fraga M, Shabafrouz K, Ribi C, Cairoli A, Guex-Crosier Y, Kuntzer T, Michielin O, Peters S, Coukos G, Spertini F, Thompson JA, Obeid M. Adverse effects of immune-checkpoint inhibitors: epidemiology, management and surveillance. Nat Rev Clin Oncol. 2019 Sep;16(9):563-580. doi: 10.1038/s41571-019-0218-0. PMID 31092901
- [Background] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084